CLINICAL TRIAL: NCT04763096
Title: A Phase IV, Single Center, Open-label, Single-arm Study to Evaluate the Efficacy and Safety of the Conversion to Tacrolimus Modified Release, ADVAGRAF® After 12 Month Treatment With a Tacrolimus Stably in Liver Transplant Recipients.
Brief Title: Evaluate the Efficacy and Safety of the ADVAGRAF®
Acronym: STABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Linical Korea (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STABLE
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Evidence of Liver Transplantation
Keywords: ADVGRAF®, Liver transplantation, tacrolimus.
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tacrolimus (Experimental): conversion to Advagraf
  Interventions: Drug: Advagraf

INTERVENTIONS:
Drug: Advagraf — Researchers must check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 5~10ng/ml of study treatment. Duration of treatment The investigational product will be administered for 24 weeks. (The lowest blood levels shall be adjusted at the discretion of the researchers, taking a blood sample is carried out in the morning before administrated of Investigational Product)
  Tacrolimus blood level is 3-10 ng/ml for 6 months prior to screening and during the maintenance therapy.
  ( ① -1day to enrollment : swich to the day before ADVAGRAF®, ② 0day to enrollment : the day swich to ADVAGRAF® )
  Duration of treatment the investigational product will be administered for 24 weeks.
  Other Names: tacrolimus

SUMMARY:
The primary objective of this study is to evaluate the efficacy of 6-month treatment with Advagraf® converted from 12-month treatment with tacrolimus in stable liver transplant recipients.

The secondary objective of this study is to evaluate severity of acute rejection confirmed by biopsy in 24 weeks, incidence of chronic rejection, patient and graft survival rates in 24 weeks, incidence of adverse events, blood pressure, tacrolimus trough level, drug compliance, and adherence.

DETAILED DESCRIPTION:
This is single-center, single-group, open-label study, phase 4 IIT. The Subject is transplantated liver at a minimum of 12 month of screening and at least 12 month Treatment with a Tacrolimus stably And start screening after obtain consent to participate in clinical trials, if appropriate in the selection criteria do not apply to the exclusion criteria are enrolled in clinical trials.

Administration method is following : The total daily dose of -1 tacrolimus will be converted to 1:1 (mg:mg) and the total daily dose of ADVAGRAF® will be administered only once daily in the morning for 24 weeks, starting from Day 0.

Researchers must check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 5~10ng/ml of study treatment.

Duration of treatment : The investigational product will be administered for 24 weeks.

Tacrorimus blood level is 3-10 ng/ml for 6 months prior to screening and during the maintenance therapy. It is recommended to check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 5~10ng/ml of study treatment. (The lowest blood levels shall be adjusted at the discretion of the researchers, taking a blood sample is carried out in the morning before have of Investigational Product)

Subjects, who participated in this clinical trial, are scheduled up to 5 times, and it will be proceed for 24 weeks. (screening and baseline, 3 weeks, 12 weeks, 24 weeks) admitted for 24 weeks including a screening visit.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 19 and 80 years old
2. Those who were transplantated liver at a minimum of 12 month of screening and after 12 month Treatment with a Tacrolimus stably.(Brain dead transplantation or biological transplant no values)
3. tacrolimus blood everage level is 3-10 ng/ml for at least 6 months prior to screening.
4. Female subjects of child bearing potential must have a negative urine or serum pregnancy test prior to enrollment and at the end of study and must agree to practice effective birth control during the study.
5. Subjects are stable clinically in the opinion of the investigator.
6. Subjects capable of understanding the purpose and risks of the study, having been fully informed and has given written informed consent to participate in the study

Exclusion Criteria:

1. Subjects having previously received an organ transplant excluding liver transplant. Or Subjects receiving an auxiliary graft or in whom a bio-artificial liver(cell system) has been used.
2. Acute rejection confirmed by histologic response or the patient had chronic rejection
3. Subjects diagnosed new malignant tumor before the pre-screening within five years , with the exception of basalioma or squamous cell carcinoma or carcinoma in situ of the skin that has been treated successfully.
4. Subjects allergic to tacrolimus or investigational product.
5. Subjects are unstable clinically state in the opinion of the investigator.
6. Subjects with any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator.
7. Subjects participating or having participated in another clinical trial and/or those taking or having taken an investigational / non-registered drug in the past 28 days.
8. Subjects taking forbidden concomitant medications or within 28 days prior to enroll.
9. Subjects who are pregnant or breast-feeding mother.
10. Subjects unlikely to comply with the visits scheduled in the protocol.
11. Subjects with renal dysfunction on the investigator's point of view or serum creatinine > 1.6mg/dL or GFR(MDRD)<30mL/min in the baseline.
12. Hepatic dysfunction: rising more than double the normal range of SGPT/ALT and/or SGOT/AST and/or bilirubin, hepatic cirrhosis

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Incidence of acute rejection confirmed by biopsy in 24 weeks after conversion | within 24 weeks
  * Incidence of acute rejection (%) = no. of subjects who had acute rejection at least once / no. of all the subjects in the relevant analysis set * 100
  * Only acute rejection confirmed by biopsy will be recognized.
  * In addition, concomitant immunosuppressants other than tacrolimus will be divided into sub-groups (by type and dosage/administration), and point estimation and calculation of 95% two-sided confidence interval will be conducted for incidence of acute rejection.

SECONDARY OUTCOMES:
Severity of acute rejection confirmed by biopsy in 24 weeks after conversion | within 24 weeks
  * For the subjects who developed acute rejection at least once, severity of acute rejection is defined as the highest severity.
Incidence of chronic rejection | within 24 weeks
  * Chronic rejection will be confirmed by biopsy.
Patient and graft survival rates in 24 weeks after conversion | within 24 weeks
Time from conversion to onset of acute rejection | within 24 weeks
Tacrolimus trough level at each visit | within 24 weeks
Incidence of adverse events | within 24 weeks
Tacrolimus compliance | within 24 weeks
  Evaluation of adherence through a subject questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ki Won Song, doctral, Principal Investigator — Asan Medical Center, Hepatobiliary, Liver Transplantion Surgery center
Locations (1):
- Seoul Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Bunzel B, Laederach-Hofmann K. Solid organ transplantation: are there predictors for posttransplant noncompliance? A literature overview. Transplantation. 2000 Sep 15;70(5):711-6. doi: 10.1097/00007890-200009150-00001. PMID 11003346
- [Result] Laederach-Hofmann K, Bunzel B. Noncompliance in organ transplant recipients: a literature review. Gen Hosp Psychiatry. 2000 Nov-Dec;22(6):412-24. doi: 10.1016/s0163-8343(00)00098-0. PMID 11072057
- [Result] Schweizer RT, Rovelli M, Palmeri D, Vossler E, Hull D, Bartus S. Noncompliance in organ transplant recipients. Transplantation. 1990 Feb;49(2):374-7. doi: 10.1097/00007890-199002000-00029. PMID 2305467
- [Result] Jain AB, Kashyap R, Rakela J, Starzl TE, Fung JJ. Primary adult liver transplantation under tacrolimus: more than 90 months actual follow-up survival and adverse events. Liver Transpl Surg. 1999 Mar;5(2):144-50. doi: 10.1002/lt.500050209. PMID 10071354
- [Result] Dopazo C, Rodriguez R, Llado L, Calatayud D, Castells L, Ramos E, Molina V, Garcia R, Fabregat J, Charco R. Successful conversion from twice-daily to once-daily tacrolimus in liver transplantation: observational multicenter study. Clin Transplant. 2012 Jan-Feb;26(1):E32-7. doi: 10.1111/j.1399-0012.2011.01521.x. Epub 2011 Sep 30. PMID 21958123
- [Result] Trunecka P, Boillot O, Seehofer D, Pinna AD, Fischer L, Ericzon BG, Troisi RI, Baccarani U, Ortiz de Urbina J, Wall W; Tacrolimus Prolonged Release Liver Study Group. Once-daily prolonged-release tacrolimus (ADVAGRAF) versus twice-daily tacrolimus (PROGRAF) in liver transplantation. Am J Transplant. 2010 Oct;10(10):2313-23. doi: 10.1111/j.1600-6143.2010.03255.x. Epub 2010 Sep 14. PMID 20840481
- [Result] Comuzzi C, Lorenzin D, Rossetto A, Faraci MG, Nicolini D, Garelli P, Bresadola V, Toniutto P, Soardo G, Baroni GS, Adani GL, Risaliti A, Baccarani U. Safety of conversion from twice-daily tacrolimus (Prograf) to once-daily prolonged-release tacrolimus (Advagraf) in stable liver transplant recipients. Transplant Proc. 2010 May;42(4):1320-1. doi: 10.1016/j.transproceed.2010.03.106. PMID 20534291
- [Result] Merli M, Di Menna S, Giusto M, Giannelli V, Lucidi C, Loria I, Ginanni Corradini S, Mennini G, Rossi M. Conversion from twice-daily to once-daily tacrolimus administration in liver transplant patient. Transplant Proc. 2010 May;42(4):1322-4. doi: 10.1016/j.transproceed.2010.04.012. PMID 20534292
- [Result] Marin-Gomez LM, Gomez-Bravo MA, Alamo-Martinez JA, Barrera-Pulido L, Bernal Bellido C, Suarez Artacho G, Pascasio JM. Evaluation of clinical safety of conversion to Advagraf therapy in liver transplant recipients: observational study. Transplant Proc. 2009 Jul-Aug;41(6):2184-6. doi: 10.1016/j.transproceed.2009.06.085. PMID 19715867
- [Result] Kim SH, Lee SD, Kim YK, Park SJ. Conversion of twice-daily to once-daily tacrolimus is safe in stable adult living donor liver transplant recipients. Hepatobiliary Pancreat Dis Int. 2015 Aug;14(4):374-9. doi: 10.1016/s1499-3872(15)60378-2. PMID 26256081
- See also: test link(2000 Sep 15;70(5):711-6.) — https://www.ncbi.nlm.nih.gov/pubmed/11003346
- See also: test link(2000 Nov-Dec;22(6):412-24.) — https://www.ncbi.nlm.nih.gov/pubmed/11072057
- See also: test link(1990 Feb;49(2):374-7.) — https://www.ncbi.nlm.nih.gov/pubmed/2305467
- See also: test link(1999 Mar;5(2):144-50.) — https://www.ncbi.nlm.nih.gov/pubmed/10071354
- See also: test link(2012 Jan-Feb;26(1):E32-7. doi: 10.1111/j.1399-0012.2011.01521.x. Epub 2011 Sep 30.) — https://www.ncbi.nlm.nih.gov/pubmed/21958123
- See also: test link(2010 Oct;10(10):2313-23. doi: 10.1111/j.1600-6143.2010.03255.x. Epub 2010 Sep 14.) — https://www.ncbi.nlm.nih.gov/pubmed/20840481
- See also: test link( 2010 May;42(4):1320-1. doi: 10.1016/j.transproceed.2010.03.106.) — https://www.ncbi.nlm.nih.gov/pubmed/20534291
- See also: test link(2010 May;42(4):1322-4. doi: 10.1016/j.transproceed.2010.04.012.) — https://www.ncbi.nlm.nih.gov/pubmed/20534292
- See also: test link(2009 Jul-Aug;41(6):2184-6. doi: 10.1016/j.transproceed.2009.06.085.) — https://www.ncbi.nlm.nih.gov/pubmed/19715867
- See also: test link(2015 Aug;14(4):374-9.) — https://www.ncbi.nlm.nih.gov/pubmed/26256081